CLINICAL TRIAL: NCT02193048
Title: Prospective Evaluation of a Scoring System in Patients Newly Diagnosed With Crohn's Disease
Acronym: PROGNOS
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000150
Record Dates: First submitted 2014-07-16; First posted 2014-07-17 (Estimated); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients newly diagnosed with Crohn's disease: This study will evaluate a new clinical scoring system in patients receiving routine treatment
  Interventions: Other: This study will evaluate a new clinical scoring system in patients receiving routine treatment

INTERVENTIONS:
Other: This study will evaluate a new clinical scoring system in patients receiving routine treatment — Treatment for Crohn's disease will be performed routinely based on the treating physicians clinical determination and patients' needs.

SUMMARY:
The purpose of this study is to prospectively evaluate a scoring system to predict a mild course of disease in patients newly diagnosed with Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

All patients with Crohn's disease who

* have been newly diagnosed (initial diagnosis not more than 6 weeks previously) and
* are as yet untreated (permitted medications are a maximum of 10 days of 5-aminosalicylates (5-ASA) or glucocorticosteroids and antibiotics for non-intestinal indications) and
* have consented to the documentation of their patient data and
* agree to the up to 5-year documentation of the course of disease

Exclusion Criteria:

* Pre-treatment with 5-ASA > 10 days
* Treatment with steroids > 10 days
* Treatment with antibiotics, immunosuppressants or biological agents > 10 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specialist gastroenterological centres
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2014-09; Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of a Crohn's scoring system | Up to 5 years
  Measured as percentage of patients with a low score at initial diagnosis having a mild course of disease during the 5 year follow-up period.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (1):
- Investigational site (there may be other sites in this country), Altenholz, Germany

REFERENCES:
- [Result] Kruis W, Bokemeyer B, Jessen P, Hoesl M, Mross M, Morgenstern J, Reimers B, Muller-Grage N, Leifeld L. Prospective Evaluation of the Prediction Score for a Mild Course of Crohn's Disease (PreMiCC) in Newly Diagnosed Patients With Crohn's Disease: The PROGNOS Study. Inflamm Bowel Dis. 2025 Mar 3;31(3):677-685. doi: 10.1093/ibd/izae086. PMID 38648264